CLINICAL TRIAL: NCT03108352
Title: Multi-center, Randomized, Double-masked, Placebo-controlled Phase III Clinical Study of Conbercept Ophthalmic Injection for Patients With BRVO.
Brief Title: Conbercept Ophthalmic Injection for Patients With Macular Edema Caused by Branch Retinal Vein Occlusion
Acronym: BRAVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chengdu Kanghong Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KH902-BRVO-CRP-1.0
Record Dates: First submitted 2017-02-08; First posted 2017-04-11 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Branch Retinal Vein Occlusion; Macular Edema
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conbercept ophthalmic injection (Experimental): Conbercept ophthalmic injection
  Interventions: Drug: Conbercept ophthalmic injection
- Sham Comparator (Sham Comparator): sham / Conbercept ophthalmic injection
  Interventions: Drug: Conbercept ophthalmic injection; Other: sham/Conbercept ophthalmic injection

INTERVENTIONS:
Drug: Conbercept ophthalmic injection — Conbercept ophthalmic injection at a dose of 0.5 mg every month(day0-month 5); If sbujects meets the criteria for repeated administration, the subject receives 0.5 mg Conbercept injection into the study eye (Month 6 ~ 11)
Other: sham/Conbercept ophthalmic injection — Sham injection every month (Day 0 - Month 5); 0.5 mg Conbercept ophthalmic injection in month 6; If sbujects meets the criteria for repeated administration, the subject receives 0.5 mg Conbercept injection into the study eye (Month 7 ~ 11)
  Arms: Sham Comparator

SUMMARY:
The purpose of this study is to verify the efficacy and safety of intravitreal injection of conbercept in patients with macular edema (ME) caused by branch retinal vein occlusion (BRVO).

ELIGIBILITY:
Inclusion Criteria:

* Patients have signed informed consent form and agreed to be followed up as per the trial protocol;
* Aged ≥ 18 years, male or female;
* Study eyes must meet all of following requirements:

  * Suffering from macular edema secondary to BRVO that involves the fovea and BRVO has been first diagnosed within previous 12 months;
  * Best corrected visual acuity (BCVA) ≥24 and ≤73 letters (Snellen equivalent is 20/320 - 20/40);
  * Central retinal thickness (CRT) on OCT is ≥300 μm;
* Without opacities in the refractive media and pupillary miosis that affects fundus examination.

Note: The eye of interest is determined by the researcher from a medical point of view if both eyes of the patient meet the inclusion criteria. In principle, the eye with poor eyesight or thicker central retina should be selected as the eye of interest.

Exclusion Criteria:

Any subject who has any of the following ocular condition:

1. Eye of interest

   * Has active retina and/or iris neovascularization;
   * Has macular epiretinal membranes or vitreous tractions which are considered to influence the central visual acuity by the researcher;
   * Has other diseases which are considered to influence the macular functional recovery by the researcher, e.g., foveal atrophy, subfoveal hemorrhage, macular hard exudates or dense submacular hard exudates;
   * Has a history of any type of retinal detachment;
   * Has non-RVO ocular diseases which are considered to possibly cause macular edema, declined visual acuity or retinal neovascularization during the study period by the researcher, e.g., wet AMD, diabetic retinopathy, uveitis/other intraocular inflammatory diseases, neovascular glaucoma and cystoid macular edema;
   * Is considered to require cataract surgery in the next 12 months by the researcher;
   * Has received intravitreal injection of corticosteroids within three months before screening, subconjunctival injection of corticosteroids within six months, or local treatment with ocular corticosteroids within one month;
   * Has received the following ophthalmic operations: scleral buckling, verteporfin-photodynamic therapy (PDT), vitrectomy, radial optic neurotomy/optic nerve sheathotomy, glaucoma filtration, parafoveal laser photocoagulation, pan-retinal photocoagulation, and macular translocation;
   * Has received YAG laser treatment or any other ophthalmic treatments (including cataract surgery, macular grid laser photocoagulation, local retinal photocoagulation, and keratoplasty) within three months before screening;
   * Has a BCVA increment by more than 10 alphabets during the screening period (BCVA tested within 24 hours before medication at Day 0 versus BCVA at the time of screening);
   * Has aphakic eye (excluding pseudophakic) or or posterior lens capsule (except YAG laser posterior capsulotomy after intraocular lens implantation);
2. Either eye:

   * Has active periocular or ocular inflammation (e.g., blepharitis, infective conjunctivitis, keratitis, scleritis, uveitis, and endophthalmitis);
   * Has previous or existing uncontrollable glaucoma (defined as IOP remaining at ≥ 30 mmHg after anti-glaucoma treatment), or has a cup-to-disc ratio of the eye of interest of above 0.8 due to severe glaucoma;
   * Has received intravitreal injection of any anti-VEGF agents (e.g.,ranibizumab, bevacizumab, and conbercept) within three months before screening;

Patient with any of the following systemic diseases:

* Has a history of anaphylaxis and allergy to fluorescein sodium, and of allergy to protein products for diagnosis or treatment, and is allergic to no less than two drugs and/or non-drug factors, or suffers from allergic diseases now;
* Has a history of stroke, has a history of myocardial and/or cerebral infarction(s) and of transient cerebral ischemia within 6 months before screening, and has active and disseminated intravascular coagulation and distinct bleeding tendency;
* Has confirmed systemic immune disease (e.g., ankylosing spondylitis, systemic lupus erythematosus, and Behcet's disease, rheumatoid arthritis, and scleroderma);
* Has any uncontrollable clinical problem (e.g., AIDS, active hepatitis, severe mental, neurological, cardiovascular and respiratory diseases, and malignancies);
* Hyperpietics with poor blood pressure control (defined as SBP remaining at ≥ 160 mmHg or DBP remaining ≥ 100 mmHg after antihypertensives therapy);
* Has a surgical history within one month before screening, and/or has unhealed wounds, ulcers and fractures at present;
* Has systemically used corticosteroids (orally, intramuscularly, intravenously) within 6 months before screening;
* Has received systemic treatment with anti-VEGF agent(s) (e.g., bevacizumab) within 6 months before screening; Patients with any of the following abnormal laboratory tests
* Those who have hepatic, renal and immunologic dysfunction (this trial specifies that ALT and AST are twice as high as the ULN of this central laboratory, and that Crea and BUN are 1.5-fold as high as the ULN of this central laboratory);
* Those who have coagulation abnormalities (PT is 3 seconds greater than or equal to the ULN, and APTT is 10 seconds greater than or equal to the ULN); Patients of childbearing age with any of the following condition
* Those who do not take effective contraceptive measures at childbearing age; Note: The following conditions are not included in the exclusion range.

  1. Amenorrhea for 12 months under the natural condition, or amenorrhea for 6 months under the natural condition and the serum FSH level of < 40 mIU/ml;
  2. Six weeks after bilateral ovariectomy with/without hysterectomy;
  3. Use of the following one or more acceptable contraceptions:

     * Sterilization (for males, with bilateral vasoligation and vasectomy)
     * Hormonal contraception (implantable, patchable, oral)
     * Intrauterine device and dural barrier method
  4. Ability to take reliable contraceptive measures over the study period and hold on to 30 days after study drug withdrawal (unacceptable contraceptive methods include: periodic continence - according to the calendar and ovulatory phase, body thermometry, post-ovulatory method, and coitus interruptus);
* Pregnant women and breastfeeding mothers (in this trial pregnancy is defined as positive U-HCG); Others
* Patient has participated in any drug (not including vitamins and minerals) clinical trial three months before screening (if the study drug has a long half-life, i.e., its five half-lives exceed three months, then it is deemed as five half-lives); Any condition in which the researcher deems necessary to be excluded in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2016-04-13 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | month 6
  Compare mean changes in Best Corrected Visual Acuity (BCVA) from baseline between the Conbercept ophthalmic injection treatment group (treatment group) and the control group at month 6.

SECONDARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) | month 3 and month 12
  1>o evaluate mean changes in BCVA from baseline of the treatment group and the control group at month 3 and 12.
Central Retinal Thickness | month 3, month 6 and month 12
  To evaluate mean changes in Central Retinal Thickness (CRT) from baseline of the treatment group and the control group at month 3, 6 and 12.
resue treament | month 6 and month 12
  To evaluate the number of subjects who received laser rescue treatment of the treatment group and the control group at month 6 and 12.
Number of participants with treatment-related the systemic and ocular safely as assessed | up to 12.5 months
  To evaluate the systemic and ocular safety of the treatment group and the control group.
distribution of BCVA changes | month 3, month 6 and month 12
  To evaluate the distribution of BCVA changes from baseline of the treatment group and the control group at month 3, 6 and 12.
mean changes in BCVA | month 0,month 1,month 2,month 3,month 4,month 5,month 6,month 7,month 8,month 9,month 10,month 11 and month 12
  To evaluate mean changes in BCVA from baseline of the treatment group and the control group at every visit.
Change in image | month 0,month 1,month 2,month 3,month 4,month 5,month 6,month 7,month 8,month 9,month 10,month 11 and month 12
  To evaluate the average changes in imaging findings (e.g., CRT and total macular volume) relative to the baseline for treatment group and control group at each follow-up visit.

OTHER OUTCOMES:
Immunogenic positive response in the treatment group | baseline,month 6, month 12
  Number of participants with Treatment-Ralated positive response to anti-drug antibody（ADA）or neutralizing antibody(Nab) in the treatment group at baseline,6 and 12months.
Immunogenic positive response in the control group | baseline,month 6, month 12
  Number of participants with Treatment-Ralated positive response to anti-drug antibody（ADA）or neutralizing antibody(Nab) in thecontrol group at baseline,6 and 12months.
safety analysis of immunogenic positive response | month 12
  To analyze the safely of subjects with positive response to ADA or Nab at 12 months after treatment and number of participants with positive respone who develop anticipants immuogenic adverse events.
safety analysis of immunogenic negative response | month 12
  To analyze the safely of subjects with negative response to ADA or Nab at 12 months after treatment and number of participants with negative response who develop anticipants immuogenic adverse events.
Best Corrected Visual Acuity (BCVA) | month 12
  To analyze the BCVA for subjects with positive response to ADA or Nab at 12 months after treatment.

CONTACTS AND LOCATIONS:
Locations (31):
- China (31):
  - The General Hospital of the People's Liberation Army, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Beijing Tongren Hospital, Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The Second Hospital of Jilin University, Changchun
  - The Second Xiangya Hospital of Central South University, Changsha
  - West China Hospital Sichuan University, Chengdu
  - Army Medical Center, Chongqing
  - The Second Hospital of Dalian Medical University, Dalian
  - Zhongshan Ophthalmic Center, Sun Yat-Sen University, Guangzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - The 2nd Affiliated Hospital of Harbin Medical University, Harbin
  - The Jiangxi Provincial People's Hospital, Nanchang
  - Jiangsu Province Hospital, Nanjing
  - Nanjing First Hospital, Nanjing
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - Eye & Ent Hospital of Fudan University, Shanghai
  - Shanghai General Hospital, Shanghai
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Zhongshan Hospital, Shanghai
  - The First Hospital of China Medical University, Shenyang
  - Tianjin Medical University Eye Hospital School of Optometry & Eye Institute, Tianjin
  - Tianjin Eye Hospital, Tianjing
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi
  - Eye Hospital,WMU Zhejiang Eye Hospital, Wenzhou
  - Wuhan General Hospital of Guangzhou Military Command, Wuhan
  - Wuxi No.2 People's Hospital, Wuxi
  - The First Affiliated Hospital of Xi'An, Xi'an

REFERENCES:
- [Derived] Shalchi Z, Mahroo O, Bunce C, Mitry D. Anti-vascular endothelial growth factor for macular oedema secondary to branch retinal vein occlusion. Cochrane Database Syst Rev. 2020 Jul 7;7(7):CD009510. doi: 10.1002/14651858.CD009510.pub3. PMID 32633861